CLINICAL TRIAL: NCT03568656
Title: An Open-label Phase I/IIa Study to Evaluate the Safety and Efficacy of CCS1477 as Monotherapy and in Combination, in Patients With Advanced Solid/Metastatic Tumours.
Brief Title: Study to Evaluate CCS1477 in Advanced Tumours
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CellCentric Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CCS1477-01
Record Dates: First submitted 2018-06-04; First posted 2018-06-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer; Metastatic Breast Cancer; Non-small Cell Lung Cancer; Advanced Solid Tumors
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — CCS1477; Abiraterone Acetate; enzalutamide; darolutamide; olaparib; atezolizumab

STUDY DESIGN:
Intervention Model Description: The RP2D/MTD dose will be determined in Part A. Parts B-H will run in parallel after the completion of Part A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- CCS1477 dose escalation - mCRPC (Experimental): CCS1477 monotherapy in patients with mCRPC
  Interventions: Drug: CCS1477
- CCS1477 expansion phase - mCRPC (Experimental): CCS1477 monotherapy in patients with mCRPC
  Interventions: Drug: CCS1477
- CCS1477 and abiraterone acetate, combination dose finding and expansion - mCRPC (Experimental): CCS1477 plus abiraterone acetate in patients with mCRPC
  Interventions: Drug: CCS1477; Drug: Abiraterone acetate
- CCS1477 and enzalutamide, combination dose finding and expansion - mCRPC (Experimental): CCS1477 plus enzalutamide in patients with mCRPC
  Interventions: Drug: CCS1477; Drug: Enzalutamide
- CCS1477 Monotherapy - Solid tumours (Experimental): CCS1477 expansion phase in patients with advanced solid tumours with molecular markers which may indicate potential for response to p300/CBP inhibition
  Interventions: Drug: CCS1477
- CCS1477 and darolutamide, combination dose finding and expansion - mCRPC (Experimental): CCS1477 plus darolutamide in patients with mCRPC
  Interventions: Drug: CCS1477; Drug: Darolutamide
- CCS1477 and olaparib, combination dose finding and expansion - mCRPC and metastatic breast cancer (Experimental): CCS1477 plus olaparib in patients with mCRPC or metastatic breast cancer.
  Interventions: Drug: CCS1477; Drug: Olaparib
- CCS1477 and atezolizumab, combination dose finding and expansion - non-small cell lung cancer (Experimental): CCS1477 plus atezolizumab in patients with non-small cell lung cancer
  Interventions: Drug: CCS1477; Drug: Atezolizumab

INTERVENTIONS:
Drug: CCS1477 — Capsules, oral
Drug: Abiraterone acetate — Abiraterone acetate 500mg tablets plus prednisone/prednisolone
  Arms: CCS1477 and abiraterone acetate, combination dose finding and expansion - mCRPC
Drug: Enzalutamide — Enzalutamide 40mg capsules/tablets
  Arms: CCS1477 and enzalutamide, combination dose finding and expansion - mCRPC
Drug: Darolutamide — 300mg tablets
  Arms: CCS1477 and darolutamide, combination dose finding and expansion - mCRPC
Drug: Olaparib — 150mg tablets
  Arms: CCS1477 and olaparib, combination dose finding and expansion - mCRPC and metastatic breast cancer
Drug: Atezolizumab — 840mg/14ml concentrate for solution for infusion vials
  Arms: CCS1477 and atezolizumab, combination dose finding and expansion - non-small cell lung cancer

SUMMARY:
A Phase 1/2a study to assess the safety, tolerability, PK and biological activity of CCS1477 in patients with metastatic castration resistant prostate cancer, metastatic breast cancer, non-small cell lung cancer or advanced solid tumours.

ELIGIBILITY:
Inclusion Criteria:

* Provision of consent
* ECOG performance status 0-1
* Assessable disease (by CT, MRI, bone scan or X-ray)
* Adequate organ function
* Highly effective contraception measures for duration of study

Additional inclusion criteria for mCRPC patients only:

* Previously received abiraterone and/or enzalutamide (or equivalent anti-androgen), and docetaxel (unless ineligible or refused)
* Progressive disease documented by one or more of the following:

  * Biochemical progression defined as at least 2 stepwise increases in a series of any 3 PSA values
  * Progression as defined by RECIST v1.1 guideline for assessment of malignant soft tissue disease.
  * Progression defined as two or more new metastatic bone lesions confirmed on bone scan from a previous assessment
* PSA at screening ≥2 μg/L
* Serum testosterone concentration ≤50 ng/dL
* Serum albumin >2.5 g/dL

Additional inclusion criteria for patients in CCS1477 plus abiraterone combination arm:

* Patients must have previously progressed on abiraterone treatment
* Patients whose last dose of abiraterone is greater than 6 months prior to start of study treatment will receive a 4-week run-in treatment with abiraterone to confirm refractoriness to abiraterone treatment

Additional inclusion criteria for patients in CCS1477 plus enzalutamide combination arm:

* Patients must have previously progressed on enzalutamide treatment
* Patients whose last dose of enzalutamide is greater than 6 months prior to start of study treatment will receive a 4-week run-in treatment with enzalutamide to confirm refractoriness to enzalutamide treatment

Additional inclusion criteria for patients in mutation arm:

* Advanced solid tumour with identification of markers which may indicate potential for response to p300/CBP inhibition. Markers include loss of function mutations in CREBBP, EP300 or ARID1A, MYC gene amplifications or rearrangements and androgen receptor (AR) gene amplifications or over-expression.

Exclusion Criteria:

* Intervention with any chemotherapy, investigational agents or other anti-cancer drugs within 14 days or 5 half-lives of the first dose
* Radiotherapy with a wide field of radiation or to more than 30% of the bone marrow within 4 weeks of the first dose of study treatment
* Major surgical procedure or significant traumatic injury within 4 weeks of the first dose of study treatment
* Strong inhibitors of CYP3A4 or CYP3A4 substrates with a narrow therapeutic range taken within 2 weeks of the first dose of study treatment
* Strong inducers of CYP3A4 within 4 weeks of the first dose of study treatment
* Statins; patients should discontinue statins prior to starting study treatment
* Any unresolved reversible toxicities from prior therapy >CTCAE grade 1 at the time of starting study treatment
* Any evidence of severe or uncontrolled systemic diseases
* Any known uncontrolled inter-current illness
* QTcF prolongation (> 480 msec).
* Primary brain tumours or known or suspected brain metastases.

Additional exclusion criteria for patients in CCS1477 plus abiraterone combination arm:

* Clinically significant cardiac abnormalities

Additional exclusion criteria for patients in CCS1477 plus enzalutamide combination arm:

* History of seizures or other predisposing factors
* Use of substrates with a narrow therapeutic index metabolised by CYP2C9 or CYP2C19 within 2 weeks of the first dose of study treatment
* Clinically significant cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2025-07-06 (Actual); Study Completion 2025-07-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | Up to 12 months
  Treatment-related adverse events and serious adverse events
Laboratory assessments | Up to 12 months
  Clinical chemistry and haematology assessments

SECONDARY OUTCOMES:
PSA response | Up to 12 months
  PSA response as defined by Prostate Cancer Clinical Trial Working Group 3 (PCWG-3)
CTC response | Up to 12 months
  CTC response defined as a change from unfavourable (five or more cells) at baseline to favourable (four or fewer cells) post treatment
Objective response rate (ORR) | Up to 12 months
  * malignant soft tissue response rate (Response Evaluation Criteria in Solid Tumours [RECIST] v1.1)
  * metastatic bone disease status (PCWG-3 bone scan criteria)
Radiological progression-free survival (rPFS) | Up to 12 months
  Defined as the time from start of treatment until objective disease progression as defined by RECIST 1.1 or PCWG-3 or death
AUC of CCS1477 | Up to 30 days after first dose of CCS1477
  Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable concentration of CCS1477
Cmax of CCS1477 | Up to 30 days after first dose of CCS1477
  Maximum observed plasma concentration (Cmax) of CCS1477

CONTACTS AND LOCATIONS:
Overall Officials: Johann de Bono, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (19):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
- France (3):
  - Institute Bergonie, Bordeaux
  - Hôpital Europeen Georges Pompidou, Paris
  - Institute Gustave Roussy, Villejuif
- Netherlands Cancer Institute (NKI), Amsterdam, Netherlands
- Spain (2):
  - Hospital Vall d'Hebron, VHIO, Barcelona
  - START CIOCC Hospital Universitario HM, Madrid
- Karolinska Institute, Stockholm, Sweden
- United Kingdom (10):
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital Cancer Centre, Birmingham
  - Cambridge University Hospital, Cambridge
  - Edinburgh Cancer Centre Western General Hospital, Edinburgh
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Leicester Royal Infirmary, Leicester
  - The Christie Hospital, Manchester
  - Freeman Hospital, Newcastle
  - University Hospital Southampton, Southampton
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caligiuri M, Williams GL, Castro J, Battalagine L, Wilker E, Yao L, Schiller S, Toms A, Li P, Pardo E, Graves B, Azofeifa J, Chicas A, Herbertz T, Lai M, Basken J, Wood KW, Xu Q, Guichard SM. FT-6876, a Potent and Selective Inhibitor of CBP/p300, is Active in Preclinical Models of Androgen Receptor-Positive Breast Cancer. Target Oncol. 2023 Mar;18(2):269-285. doi: 10.1007/s11523-023-00949-7. Epub 2023 Feb 24. PMID 36826464
- [Derived] Eickhoff N, Bergman AM, Zwart W. Homing in on a Moving Target: Androgen Receptor Cistromic Plasticity in Prostate Cancer. Endocrinology. 2022 Oct 11;163(11):bqac153. doi: 10.1210/endocr/bqac153. PMID 36125208